CLINICAL TRIAL: NCT06492408
Title: Phase II Study of Neoadjuvant CT-Guided Intra-tumor Double Checkpoint Blockades for Untreated Hepatocellular Carcinoma (HCC) Amenable for Surgical Resection
Brief Title: Neoadjuvant Intra-tumor Double Immunotherapy for Hepatocellular Carcinoma.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZ-IT-ICIs-HCC-Neoadjuvant-027
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Hepatic Cancer; Surgery
Keywords: Hepatocellular Carcinoma;; Intra-tumor injection; Neoadjuvant therapy; Surgery; Immunotherapy; CTLA4 antibody; PD1 antibody; PDL1 antibody
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Ipilimumab; pembrolizumab; durvalumab; Idarubicin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: IT injection of double ICIs (Experimental): Neoadjuvant therapy: intra-tumor injection of double ICIs only.
  Interventions: Drug: ipilimumab, pembrolizumab, durvalumab, idarubicin, bevacizumab
- Group 2: IT injection of double ICIs and chemodrug (Experimental): Neoadjuvant therapy: intra-tumor injection of double ICIs and chemodrug.
  Interventions: Drug: ipilimumab, pembrolizumab, durvalumab, idarubicin, bevacizumab
- Group 3: IT injection of double ICIs and chemodrug plus bevacizumab (Experimental): Neoadjuvant therapy: intra-tumor injection of double ICIs and chemodrug plus bevacizumab.
  Interventions: Drug: ipilimumab, pembrolizumab, durvalumab, idarubicin, bevacizumab

INTERVENTIONS:
Drug: ipilimumab, pembrolizumab, durvalumab, idarubicin, bevacizumab — This study has 3 subgroups:
  Arm 1. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab is administrated with a total dose of 1-2mg/kg via intra-tumor fine needle injection in 10 min, every 3 weeks, total 3-4 times.
  Arm 2. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab combined with idarubicin is administrated via intra-tumor fine needle injection in 15 min, every 3 weeks, total 3-4 times.
  Arm 3. Ipilimumab +pembrolizumab or Ipilimumab +durvalumab combined with idarubicin plus bevacizumab is administrated via intra-tumor fine needle injection in 20 min, every 3 weeks, total 3-4 times.
  Other Names: Other ICIs

SUMMARY:
This trial is designed to investigate the safety, response rates and survival outcomes of patients with hepatocellular carcinoma by delivery of CTLA4 and PD1 or PDL1 antibodies combination through CT-guided intra-tumor (IT) injection.

DETAILED DESCRIPTION:
Antibodies against CTLA4, PD1 or PDL1 are representative drugs for the check-points inhibitory agents, and their clinical indications have been approved in various types of tumors, including advanced melanoma, non-small cell lung cancer, renal cell carcinoma, and classical Hodgkin's lymphoma and late recurrent head and neck squamous cell carcinoma patients, et al. Those drugs are regularly systemically administrated by vein infusion, however, local delivery of those drugs via interventional radiology technique including trans-artery or intra-tumor injection may increase the local drug concentration of the tumor, improve the efficacy, and reduce systemic adverse reactions. CTLA4 antibody ipilimumab has been widely effectively using to combine with PD1 or PDL1 antibody and this study is to combine ipilimumab and PD1 antibody or PDL1 antibody, so called double checkpoint inhibitors combination therapy, as neoadjuvant therapy for hepatocellular carcinoma (HCC) via intra-tumor admistration. To the investigator's knowledge, no studies have been developed on the safety, efficacy and survival benefit of the double checkpoint inhibitors combination therapy for cancer patients as neoadjuvant treatment via intra-tumor delivery. This phase II clinical trial is designed to assess the safety and survival benefit of ipilimumab and pembrolizumab or durvalumab combination with or without chemodrug or bevacizumab as neoaduvant therapy on patients with HCC, including safety, pCR, mPR, PFS, ORR, DCR, and median survival time.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed previously untreated hepatocellular carcinoma (HCC). If a diagnostic biopsy is available, a pre-treatment biopsy is not required. Patients with a suspected HCC are eligible, but pathology must be confirmed prior to initiating treatment on study.
2. The patient must be a suitable candidate for surgery, in the opinion of the treating physician.
3. Signed and dated written informed consent must be provided by the patient prior to admission to the study in accordance with International Conference on Harmonization-Good Clinical Practice (ICH-GCP) guidelines and to the local legislation.
4. Eastern Cooperative Oncology Group (ECOG) performance status score 0-1
5. Absolute neutrophil count (ANC) >= 1.5 x 10^9/L; Hemoglobin >= 8.0 g/dL; Platelets >= 100 x 10^9/L; Total bilirubin =< 1.5 x upper limit of normal (ULN) (except subjects with Gilbert syndrome who can have total bilirubin < 3.0 mg/dL); Creatinine =< 1.5 x ULN or calculated creatinine clearance >= 50 mL/min using Cockcroft-Gault formula for creatinine clearance calculation OR 24-hour urine creatinine clearance >= 50 mL/min.
6. Birth control.
7. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Patients participated in clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
2. Patients accompany by ascites, hepatic encephalopathy and esophageal and gastric varices bleeding;
3. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
4. Patients accompanied with other tumors or past medical history of malignancy;
5. Pregnant or lactating patients, all patients participating in this trial must adopt appropriate birth control measures during treatment;
6. Patients have poor compliance. A.Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).

   B.Renal failure / insufficiency requiring hemo-or peritoneal dialysis. C.Known severe atheromatosis. D.Known uncontrolled blood hypertension (> 160/100 mm/Hg).
7. Allergic to contrast agent;
8. Any agents which could affect the absorption or pharmacokinetics of the study drugs
9. Other conditions that investigator decides not suitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate for the study groups | Six months
  Pathologic complete response (pCR) is defined as after neoadjuvant therapy, the surgical specimen can not find any residual cancer cells.
mPR rate for the study groups | Six months
  Major pathologic response (MPR) is defined as pathological less than 10% survival cancer cells after tumor resection.

SECONDARY OUTCOMES:
Toxicity of the study groups | Six months
  Toxicity is assessed by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4.
Response rates to neoadjuvant treatment | Six years
  Response rates are assessed by Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1.
Recurrence-free survival | Six years
  Recurrence-free survival is measured as routine.
Overall survival | Six years
  To correlate major pathologic response with recurrence-free and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong, China